CLINICAL TRIAL: NCT04476264
Title: Novel Use of an Adjustable Single 8-0 Polypropylene Suture of Scleral Fixation
Brief Title: Novel Use of an Adjustable Single 8-0 Polypropylene Suture of Scleral Fixation Without Conjunctival Dissection
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TR2019IOL
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Suture, Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- transscleral IOL fixation: the use of a novel adjustable single 8-0 polypropylene suture for scleral fixation without conjunctival dissection
  Interventions: Procedure: Novel use of an adjustable single 8-0 polypropylene suture of scleral fixation without conjunctival dissection

INTERVENTIONS:
Procedure: Novel use of an adjustable single 8-0 polypropylene suture of scleral fixation without conjunctival dissection — The present study serves to describe a novel approach to utilizing a single adjustable 8-0 polypropylene suture for scleral fixation without conjunctival dissection and to evaluate safety and efficacy outcomes associated with this technique.

SUMMARY:
1. observe the effectivity of an adjustable single 8-0 polypropylene suture to scleral fix without conjunctival dissection for the treatment with aphakia or inadequate posterior capsule support.
2. observe the complication of this surgery method.

ELIGIBILITY:
Inclusion Criteria:

* Any patients who used an adjustable single 8-0 polypropylene suture of scleral fixation without conjunctival dissection could be included.

Exclusion Criteria:

* Data from patients with a < 6-month postoperative follow-up or with incomplete operative or postoperative medical records were excluded from this study. Enrolled patients had complete records pertaining to their visual acuity (VA), slit-lamp photographs, and ultrasound biomicroscope (UBM) findings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any participants who used an adjustable single 8-0 polypropylene suture of scleral fixation without conjunctival dissection could be included.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
uncorrected VA | at 3 months postoperatively
  preoperative and postoperative uncorrected VA

SECONDARY OUTCOMES:
Postoperative complications | follow up time is larger 6 month
  Postoperative complications during the follow-up

OTHER OUTCOMES:
IOL and tunnel location | at 2 months postoperatively
  IOL tunnels containing sutures were clearly visible by UBM

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mo B, Li SF. Novel use of an adjustable single 8-0 polypropylene suture of scleral fixation without conjunctival dissection. BMC Ophthalmol. 2020 Jul 25;20(1):304. doi: 10.1186/s12886-020-01558-y. PMID 32711502